CLINICAL TRIAL: NCT03733730
Title: Post Approval Study of the AcrySof® IQ ReSTOR® Toric IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILR431b-P001; P040020 (Other: FDA)
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Aphakia; Presbyopia; Astigmatism
Keywords: cataract
MeSH Terms: conditions — Aphakia; Presbyopia; Astigmatism; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Arm 1 completed prior to the initiation of Arm 2. Within each arm, IOL assignment was parallel.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): ACRYSOF IQ RESTOR Multifocal Toric IOL (+3.0 D or +2.5 D) implanted in at least one eye during cataract surgery, with implantation occurring from November 2018 through July 2020.
  Interventions: Device: ACRYSOF IQ RESTOR +3.0 Multifocal Toric IOL; Device: ACRYSOF IQ RESTOR +2.5 D Multifocal Toric IOL; Procedure: Cataract Surgery
- Cohort 2 (Experimental): ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL or ACRYSOF IQ RESTOR +2.5 D Multifocal IOL implanted in at least one eye during cataract surgery, with implantation occurring after July 2020.
  Interventions: Device: ACRYSOF IQ RESTOR +3.0 Multifocal Toric IOL; Device: ACRYSOF IQ RESTOR +2.5 D Multifocal IOL; Procedure: Cataract Surgery

INTERVENTIONS:
Device: ACRYSOF IQ RESTOR +3.0 Multifocal Toric IOL — Intraocular lens (IOL) intended for visual correction of aphakia in adult patients with and without presbyopia, who desire near, intermediate and distance vision, reduction of residual cylinder and increased spectacle independence. IOLs are implantable medical devices and are intended for long term use over the lifetime of the cataract subject.
  Other Names: Models SND1T3, SND1T4, SND1T5, and SND1T6
Device: ACRYSOF IQ RESTOR +2.5 D Multifocal Toric IOL — Intraocular lens (IOL) intended for visual correction of aphakia in adult patients with and without presbyopia, who desire near, intermediate and distance vision, reduction of residual cylinder and increased spectacle independence. IOLs are implantable medical devices and are intended for long term use over the lifetime of the cataract subject.
  Other Names: Models SV25T3, SV25T4, SV25T5, and SV25T6
  Arms: Cohort 1
Device: ACRYSOF IQ RESTOR +2.5 D Multifocal IOL — Intraocular lens (IOL) intended for visual correction of aphakia in adult patients with and without presbyopia, who desire near, intermediate and distance vision with increased spectacle independence. IOLs are implantable medical devices and are intended for long term use over the lifetime of the cataract subject.
  Other Names: Model SV25T0
  Arms: Cohort 2
Procedure: Cataract Surgery — Routine small incision cataract surgery with IOL implantation

SUMMARY:
This is a prospective, multicenter, post-approval active surveillance study. The purpose of this study is to report the rate of post-surgical intraocular inflammation (based upon a specified case definition) reported within a 180-day post-surgical period following attempted implantation of an ACRYSOF IQ RESTOR Toric or ACRYSOF IQ RESTOR IOL in the US.

DETAILED DESCRIPTION:
If a second eye will participate in the study, subjects will receive the second eye cataract surgery within 20 days of the first eye surgery. Four postoperative follow-up visits are planned to occur at 1-2 days, 7-14 days, 30-60 days, and 90-180 days, for each enrolled eye. Subject participation in this study is expected to last up to 7 months, including a total of 6 study visits for subjects implanted in one eye and up to 11 visits for subjects implanted in both eyes. Upon completion of the 180 days follow-up visit, subjects will be exited from the study.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative cataract in the study eye(s)
* Planned implantation in at least one eye with:

  * Cohort 1: An ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL (Models SND1T3, SND1T4, SND1T5 or SND1T6) or an ACRYSOF IQ RESTOR +2.5 D Multifocal Toric IOLs (Models SV25T3, SV25T4, SV25T5, and SV25T6) in accordance with the product labeling from November 2018 to July 2020
  * Cohort 2: An ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL (Models SND1T3, SND1T4, SND1T5 or SND1T6), or an ACRYSOF IQ RESTOR +2.5 D Multifocal IOL (Model SV25T0) in accordance with the product labeling after July 2020.
* Able to comprehend and sign a statement of informed consent
* Willing and able to complete all required postoperative visits
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Eyes with clinically significant ocular, including adnexa, or intraocular infection or inflammation (at the screening visit prior to surgery or on the day of surgery)
* History of any intraocular inflammation within the past 12 months (ex: uveitis, choroiditis)
* Combined procedures introducing an additional medical device during cataract surgery (ex: cataract surgery with implant of glaucoma stent)
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2449 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CRD Surgical, Study Director — Alcon Research
Locations (38):
- United States (37):
  - Trinity Research Group, Dothan, Alabama
  - Eye Doctors of Arizona, Phoenix, Arizona
  - InSight Vision Center, Fresno, California
  - Harvard Eye Associates, Laguna Hills, California
  - Wolstan Goldberg Eye Associates, Torrance, California
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - Central Florida Eye Specialists, DeLand, Florida
  - Mid Florida Eye Center, Mt. Dora, Florida
  - Newsom Eye and Laser Center, Sebring, Florida
  - SightTrust Eye Institute, Sunrise, Florida
  - Gainesville Eye Associates, Gainesville, Georgia
  - Sabates Eye Center, Leawood, Kansas
  - Durrie Vision, Overland Park, Kansas
  - Senior Health Services, Louisville, Kentucky
  - Willis-Knighton Eye Institute South, Shreveport, Louisiana
  - Chu Vision Institute, Bloomington, Minnesota
  - Associated Eye Care, Stillwater, Minnesota
  - Moyes Eye Center, Kansas City, Missouri
  - St. Louis Eye Institute, Town and Country, Missouri
  - Raymond Fong Eye Care, New York, New York
  - Seeta Eye Center, Poughkeepsie, New York
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Bergstrom Eye Research, Fargo, North Dakota
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Vision for Life, Nashville, Tennessee
  - Kleinman Evangelista Eye Center of Texas, Arlington, Texas
  - Keystone Research, Austin, Texas
  - El Paso Eye Surgeons, El Paso, Texas
  - Chu Eye Institute, Fort Worth, Texas
  - Houston Eye Associates, Houston, Texas
  - Berkeley Eye Center, Houston, Texas
  - Baylor College of Medicine Alkek Eye Center, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Vistar Eye Center, Roanoke, Virginia
  - Northwest Eye Surgeons, Seattle, Washington
- Centro Oftalmologico Metropolitano, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 37 investigative sites located in the United States and 1 investigative site located in Puerto Rico.
Pre-assignment Details: Cohort 1: Of the 478 enrolled, 25 subjects discontinued prior to attempted implantation. Cohort 2: Of the 1971 enrolled, 144 subjects discontinued prior to attempted implantation. This reporting group includes all enrolled subjects/eyes with attempted implantation (453/706 in Cohort 1) (1827/3417 in Cohort 2).
Units Other Than Participants: eyes
Groups:
- Cohort 1: ACRYSOF IQ RESTOR Multifocal Toric IOL (+3.0 D or +2.5 D) implanted in at least one eye during cataract surgery.
- Cohort 2: ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL or ACRYSOF IQ RESTOR +2.5 D Multifocal IOL implanted in at least one eye during cataract surgery.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started (All subjects/eyes with attempted implantation) | 453; 706 eyes | 1827; 3417 eyes
First Eye Attempted Implantation | 453; 453 eyes | 1827; 1827 eyes
First Eye Successful Implantation | 453; 453 eyes | 1827; 1827 eyes
Second Eye Attempted Implantation | 453; 253 eyes | 1827; 1590 eyes
Second Eye Successful Implantation | 453; 253 eyes | 1827; 1589 eyes
Safety Analysis Set | 453; 706 eyes | 1827; 3417 eyes
Completed | 451; 703 eyes | 1778; 3334 eyes
Not Completed | 2; 3 eyes | 49; 83 eyes
Not completed — Lost to Follow-up | 1 | 32
Not completed — Other | 1 | 0
Not completed — Adverse Event | 0 | 4
Not completed — Death | 0 | 5
Not completed — Withdrawal by Subject | 0 | 8

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set. Cohort 2 excluded one site (35 subjects/60 eyes) due to noncompliance with GCP as previously communicated with the FDA.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 453 | 1792 | 2245
Age, Customized [Number; unit: participants]
  Less that 65 years | 148 | 432 | 580
  Equal to or greater than 65 years | 305 | 1360 | 1665
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 1150 | 1424
  Male | 179 | 642 | 821
Race/Ethnicity, Customized [Number; unit: participants]
  White | 336 | 1387 | 1723
  Black or African American | 28 | 266 | 294
  American Indian or Alaska Native | 1 | 14 | 15
  Asian | 83 | 88 | 171
  Native Hawaiian or Other Pacific Islander | 0 | 6 | 6
  Multi-Racial | 2 | 2 | 4
  Other | 3 | 29 | 32

OUTCOME MEASURES:

1. Primary Outcome: Rate of Eyes With Post-Surgical Intraocular Inflammation - By Eye - Cohort 2
Description: Post-surgical intraocular inflammation was defined as exacerbated intraocular inflammation within 180 days after IOL implantation, indicated by greater than or equal to 3+ aqueous cell within the first 14 days post-operative, and/or greater than or equal to 2+ aqueous cell greater than 14 days and less than or equal to 60 days post-operative, and/or greater than or equal to 1+ aqueous cell greater than 60 days post-operatively or later. The event rate (per 1000 IOL implants) was calculated as "Total # of reported events / Total # of implants X 1000." No formal safety hypothesis was pre-specified for this outcome measure. This outcome measure was pre-specified for Cohort 2 only.
Time Frame: Day 90 to 180 post implantation, each eye. The second eye was implanted within 20 days of the first eye.
Population: Safety Analysis Set, minus one site (35 subjects/60 eyes) due to noncompliance with GCP as previously communicated with the FDA.
Measure: Number; unit: event rate per 1000 implants
Units Other Than Participants: eyes
Groups:
- First Eye: ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL or ACRYSOF IQ RESTOR +2.5 D Multifocal IOL implanted in first eye during cataract surgery.
- Second Eye: ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL or ACRYSOF IQ RESTOR +2.5 D Multifocal IOL implanted in second eye during cataract surgery.
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 1792 | 1565
Number analyzed (eyes) | 1792 | 1565
event rate per 1000 implants | 5.6 | 4.5

2. Primary Outcome: Rate of Eyes With Post-Surgical Intraocular Inflammation - Overall Eyes - Cohort 2
Description: as for outcome 1
Time Frame: Day 90 to 180 post implantation, each eye. The second eye was implanted within 20 days of the first eye.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event rate per 1000 implants
Units Other Than Participants: eyes
Groups:
- Overall Eyes: ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL or ACRYSOF IQ RESTOR +2.5 D Multifocal IOL implanted in at least one eye during cataract surgery.
Arm/Group | Overall Eyes
Number analyzed (Participants) | 1792
Number analyzed (eyes) | 3357
event rate per 1000 implants | 5.1 [2.95 to 8.10]

3. Secondary Outcome: Rate of Eyes With Toxic Anterior Segment Syndrome (TASS) - By Eye - Cohort 2
Description: TASS was defined as exacerbated intraocular inflammation within 180 days after IOL implantation associated with the following findings: Greater than or equal to 3+ aqueous cell, non-infectious etiology, and rapid onset (up to and including 2 days post-operatively). The event rate (per 1000 IOL implants) was calculated as "Total # of reported events / Total # of implants X 1000." No formal safety hypothesis was pre-specified for this outcome measure. This outcome measure was pre-specified for Cohort 2 only.
Time Frame: Day 90 to 180 post implantation, each eye. The second eye was implanted within 20 days of the first eye.
Population: as for outcome 1
Measure: Number; unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 1792 | 1565
Number analyzed (eyes) | 1792 | 1565
event rate per 1000 implants | 1.1 | 0.0

4. Secondary Outcome: Rate of Eyes With Toxic Anterior Segment Syndrome (TASS) - Overall Eyes - Cohort 2
Description: as for outcome 3
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | Overall Eyes
Number analyzed (Participants) | 1792
Number analyzed (eyes) | 3357
event rate per 1000 implants | 0.6 [0.07 to 2.15]

5. Secondary Outcome: Rate of Eyes With Acute Postoperative Endophthalmitis - By Eye - Cohort 2
Description: Acute postoperative endophthalmitis was defined as exacerbated intraocular inflammation within 180 days after IOL implantation associated with the following findings: Greater or equal to 3+ aqueous cell, etiology (infectious per positive culture of ocular media; non-infectious per negative culture of ocular media), inflammatory cells in the vitreous and/or vitreous abscess, and rapid onset (3 to 14 days post-operatively). The event rate (per 1000 IOL implants) was calculated as "Total # of reported events / Total # of implants X 1000." No formal safety hypothesis was pre-specified for this outcome measure. This outcome measure was pre-specified for Cohort 2 only.
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number; unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 1792 | 1565
Number analyzed (eyes) | 1792 | 1565
event rate per 1000 implants | 0.0 | 0.6

6. Secondary Outcome: Rate of Eyes With Acute Postoperative Endophthalmitis - Overall Eyes - Cohort 2
Description: as for outcome 5
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | Overall Eyes
Number analyzed (Participants) | 1792
Number analyzed (eyes) | 3357
event rate per 1000 implants | 0.3 [0.01 to 1.66]

7. Secondary Outcome: Rate of Eyes With Chronic Postoperative Endophthalmitis - By Eye - Cohort 2
Description: Chronic postoperative endophthalmitis was defined as exacerbated intraocular inflammation within 180 days after IOL implantation associated with the following findings: Greater than or equal to 1+ aqueous cell, etiology (infectious per positive culture of ocular media; non-infectious per negative culture of ocular media), inflammatory cells in the vitreous, and delayed onset (greater than 14 days post-operatively). The event rate (per 1000 IOL implants) was calculated as "Total # of reported events / Total # of implants X 1000." No formal safety hypothesis was pre-specified for this outcome measure. This outcome measure was pre-specified for Cohort 2 only.
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number; unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 1792 | 1565
Number analyzed (eyes) | 1792 | 1565
event rate per 1000 implants | 0.0 | 0.0

8. Secondary Outcome: Rate of Eyes With Chronic Postoperative Endophthalmitis - Overall Eyes - Cohort 2
Description: as for outcome 7
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | Overall Eyes
Number analyzed (Participants) | 1792
Number analyzed (eyes) | 3357
event rate per 1000 implants | 0.0 [0.00 to 1.10]

9. Secondary Outcome: Rate of Eyes With Uncategorized Cases of Post-Surgical Intraocular Inflammation - By Eye - Cohort 2
Description: Uncategorized post-surgical intraocular inflammation was defined as signs of exacerbated intraocular inflammation within 180 days after IOL implantation associated with the following findings that do not fall in the given category of TASS, Acute Postoperative Endophthalmitis, or Chronic Postoperative Endophthalmitis: Greater than or equal to 3+ aqueous cell within the first 14 days post-op, and/or greater than or equal to 2+ aqueous cell greater than 14 days and less than or equal to 60 days post-op, and/or greater than or equal to 1+ aqueous cell greater than 60 days post-operatively or later. The event rate (per 1000 IOL implants) was calculated as "Total # of reported events / Total # of implants X 1000." No formal safety hypothesis was pre-specified for this outcome measure. This outcome measure was pre-specified for Cohort 2 only.
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number; unit: event rate per 1000 implants
Units Other Than Participants: eyes
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 1792 | 1565
Number analyzed (eyes) | 1792 | 1565
event rate per 1000 implants | 4.5 | 3.8

10. Secondary Outcome: Rate of Eyes With Uncategorized Cases of Post-Surgical Intraocular Inflammation - Overall Eyes - Cohort 2
Description: as for outcome 9
Time Frame: Day 90 to 180 post second eye implantation, with the second implantation occurring up to 20 days after the first
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: event rate per 1000 implants
Units Other Than Participants: eyes
Groups:
- Overall: ACRYSOF IQ RESTOR +3.0 D Multifocal Toric IOL or ACRYSOF IQ RESTOR +2.5 D Multifocal IOL implanted in at least one eye during cataract surgery.
Arm/Group | Overall
Number analyzed (Participants) | 1792
Number analyzed (eyes) | 3357
event rate per 1000 implants | 4.2 [2.28 to 6.99]

ADVERSE EVENTS:
Time Frame: Cohort 1 and Cohort 2: Adverse events (AEs) were collected pre-treatment (Day -40 or less pre-surgery first eye) up to Day 90-180 post-surgery/study exit. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: Safety Analysis Set: All subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye). The "At Risk" population for pretreatment and systemic AEs is reported in units of subjects. The "At Risk" population for ocular AEs is reported in units of eyes. Only total subjects/eyes affected by other non-serious AEs that occurred at greater than 5% are reported.
Groups:
- Cohort 1 Pretreatment; Cohort 2 Pretreatment: Events reported in this group occurred prior to attempted implantation with the ACRYSOF IQ RESTOR Multifocal IOL
- Cohort 1 Ocular - First Eye; Cohort 2 Ocular - First Eye: Events reported in this group occurred after attempted implantation with the ACRYSOF IQ RESTOR Multifocal IOL and include ocular events in the first implanted eye
- Cohort 1 Ocular - Second Eye; Cohort 2 Ocular - Second Eye: Events reported in this group occurred after attempted implantation with the ACRYSOF IQ RESTOR Multifocal IOL and include ocular events in the second implanted eye
- Cohort 1 Systemic; Cohort 2 Systemic: Events reported in this group occurred after attempted implantation with the ACRYSOF IQ RESTOR Multifocal IOL
Arm/Group | Cohort 1 Pretreatment | Cohort 1 Ocular - First Eye | Cohort 1 Ocular - Second Eye | Cohort 1 Systemic | Cohort 2 Pretreatment | Cohort 2 Ocular - First Eye | Cohort 2 Ocular - Second Eye | Cohort 2 Systemic
All-Cause Mortality (participants affected / at risk) | 0/453 | 0/453 | 0/253 | 0/453 | 0/1827 | 0/1827 | 0/1590 | 7/1827
Serious Adverse Events (participants affected / at risk) | 0/453 | 4/453 | 6/253 | 8/453 | 5/1827 | 27/1827 | 17/1590 | 28/1827
Other Adverse Events (participants affected / at risk) | 2/453 | 71/453 | 31/253 | 0/453 | 0/1827 | 0/1827 | 0/1590 | 0/1827
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Pretreatment (N=453) | Cohort 1 Ocular - First Eye (N=453) | Cohort 1 Ocular - Second Eye (N=253) | Cohort 1 Systemic (N=453) | Cohort 2 Pretreatment (N=1827) | Cohort 2 Ocular - First Eye (N=1827) | Cohort 2 Ocular - Second Eye (N=1590) | Cohort 2 Systemic (N=1827)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Anterior capsule contraction (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Corneal infiltrates (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glare (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Refraction disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vitreoretinal traction syndrome (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous prolapse (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 6 | 4 | 0
Posterior capsule rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0 | 0 | 4 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral endovascular aneurysm repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Corneal operation (Surgical and medical procedures) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intra-ocular injection (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Intraocular lens repositioning (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0 | 7 | 4 | 0
Lens extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 0
Lung lobectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mastectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal laser coagulation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Retinal operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Retinopexy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Spinal Operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Pretreatment (N=453) | Cohort 1 Ocular - First Eye (N=453) | Cohort 1 Ocular - Second Eye (N=253) | Cohort 1 Systemic (N=453) | Cohort 2 Pretreatment (N=1827) | Cohort 2 Ocular - First Eye (N=1827) | Cohort 2 Ocular - Second Eye (N=1590) | Cohort 2 Systemic (N=1827)
Dry eye (Eye disorders) | 2 | 23 | 11 | 0 | 0 | 0 | 0 | 0
Posterior capsule opacification (Eye disorders) | 0 | 31 | 13 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 27 | 11 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT03733730/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03733730/SAP_001.pdf